CLINICAL TRIAL: NCT00667303
Title: Prospective Surveillance For Respiratory Virus Infections In Children Undergoing Hematopoietic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BMTRV
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Respiratory Virus Infections
Keywords: Hematopoietic stem cell transplant

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal washes Fluorescent antibody detection Respiratory viral culture
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: Nasopharyngeal Washes; Other: Fluorescent antibody detection; Other: Respiratory viral culture

INTERVENTIONS:
Other: Nasopharyngeal Washes — A total of eight nasopharyngeal washes will be done at the following time points: Prior to conditioning, on the day of admission and thereafter every two weeks until day +100 (Day +14, 28, 42, 56, 70, 84 and 98). To allow for flexibility over the weekends and holidays the specimen may be collected on the scheduled day ± 3 days. The baseline sample obtained prior to conditioning is required for patient to be considered evaluable.
Other: Fluorescent antibody detection — For IF (Direct IF for hHRSV and indirect IF for the other viruses), the specimens will be spotted onto glass slides. Samples without respiratory epithelial cells will be considered inconclusive. Labelled antibodies against Flu A, Flu B, HPIV 1 to 3, RSV, hMPV and Adv will be used.
Other: Respiratory viral culture — Shell vial culture specimens will be inoculated and incubated for 48 hours. The following RVs: Flu A, Flu B, HPIV 1-3, RSV, Adv and hMPV will be identified on the basis of cytopathic effects in cell cultures and confirmed by staining with fluorescein-conjugated monoclonal antibodies.

SUMMARY:
The Study aims to prospectively survey the incidence of respiratory virus infections using molecular methodologies, in children undergoing hematopoietic stem cell transplantation

DETAILED DESCRIPTION:
Samples will be collected with a nasopharyngeal wash and processed for direct fluorescent antibody, culture and Polymerase chain reaction (PCR)

ELIGIBILITY:
Inclusion Criteria:

* Age: Birth to 18 years.
* Patients undergoing an allogeneic HSCT for any disease.
* Parent or guardian willing to sign informed consent.

Exclusion Criteria:

* Intra nasal lesion which precludes the performance of the nasopharyngeal wash.
* Patients on Continuous Positive Airway Pressure (CPAP) or Bilevel Positive Airway Pressure (BiPAP).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, birth to 18 years old, within the first 100 days of a hematopoietic stem cell transplant who are either asymptomatic, or symptomatic with an upper respiratory tract infection (URTI) or a lower respiratory tract infection (LRTI).
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2007-12; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Incidence of RV infection at any time after transplant: The day of onset of an infection is defined as the day when the first positive diagnostic test was performed. | All patients will be followed until day +100 after the HSCT.

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Srinivasan, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org